CLINICAL TRIAL: NCT03452722
Title: Neuroinflammatory Response in Patients With ICH and IVH Treated With rtPA
Status: Completed | Type: Observational
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Matija Sošić, MD, University of Rijeka
Other Study IDs: 13.06.1.1.12
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hypertensive Intracerebral Hemorrhage; Intraventricular Hemorrhage; Brain Injuries
Keywords: secondary brain injury; neuroinflammation
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive; Brain Injuries; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: Applied rtPA
  Interventions: Drug: intraventricual recombinant tissue plasminogen activator application
- Control study: rtPA not applied

INTERVENTIONS:
Drug: intraventricual recombinant tissue plasminogen activator application
  Groups: Study group

SUMMARY:
This study compares the neuroinflammatory response in patients with hypertensive ICH associated with IVH treated with intraventriculary applied rtPA, and the control group. The inflammatory mediator concentration is analyzed in local cerebrospinal liquor.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with primary ICH with IVH
* ICH score 2-4, , with origin of the hematoma in the basal ganglia and blood in the third and/or ventricle
* Patient is not considered a surgical candidate by neurosurgery service

Exclusion Criteria:

* No history of diseases or drugs that affect the immunological system.
* ICH score 1 and 5
* Current participation in another research drug treatment protocol
* Previously known intracranial arteriovenous malformation or aneurysms
* Intracerebral hematoma considered to be related to trauma
* ICH is located in the pons
* Blood in the subarachnoid space visualized on CT scan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects from 18 to 80 years.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Cytokine concentration difference between two groups | Samples taken on day 0, day 1, day 3 and day 7.
  Cytokine concentration measured from CSL

CONTACTS AND LOCATIONS:
Overall Officials: Vlatka Sotosek Tokmadzic, PhD, Study Director — University of Rijeka

REFERENCES:
- [Background] Hanley DF, Lane K, McBee N, Ziai W, Tuhrim S, Lees KR, Dawson J, Gandhi D, Ullman N, Mould WA, Mayo SW, Mendelow AD, Gregson B, Butcher K, Vespa P, Wright DW, Kase CS, Carhuapoma JR, Keyl PM, Diener-West M, Muschelli J, Betz JF, Thompson CB, Sugar EA, Yenokyan G, Janis S, John S, Harnof S, Lopez GA, Aldrich EF, Harrigan MR, Ansari S, Jallo J, Caron JL, LeDoux D, Adeoye O, Zuccarello M, Adams HP Jr, Rosenblum M, Thompson RE, Awad IA; CLEAR III Investigators. Thrombolytic removal of intraventricular haemorrhage in treatment of severe stroke: results of the randomised, multicentre, multiregion, placebo-controlled CLEAR III trial. Lancet. 2017 Feb 11;389(10069):603-611. doi: 10.1016/S0140-6736(16)32410-2. Epub 2017 Jan 10. PMID 28081952
- [Background] Dunatov S, Antoncic I, Bralic M, Jurjevic A. Intraventricular thrombolysis with rt-PA in patients with intraventricular hemorrhage. Acta Neurol Scand. 2011 Nov;124(5):343-8. doi: 10.1111/j.1600-0404.2010.01481.x. Epub 2011 Feb 8. PMID 21303348